CLINICAL TRIAL: NCT00416130
Title: Phase I/II Clinical Trial of Vorinostat in Patients With Recurrent and/or Metastatic Breast Cancer
Brief Title: Clinical Trial of SAHA in Patients With Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Lee Soo Chin, National University Hospital, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR05/24/06; DSRB Reference Code: B/06/275 (Other: NHG Domain Specific Review Board); HSA No: CTC0600314 (Other: Health Science Authority (Singapore))
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: Phase I/II Clinical Trial; Vorinostat; SAHA; Recurrent Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat (Experimental): A phase I portion that will determine the safety of 400mg Vorinostat once a day, continuously in the Asian population. A pre-determined dose reduction schema will be followed in the event of significant dose-limiting toxicities at this dose. Phase II will recruit additional patients at the determined dose with the goal of evaluating drug efficacy.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — MK-0683 capsules, 100 mg, 400mg once a day, continuously (at dose level 0 - Phase 1 part of the study)
  Other Names: MK-0683

SUMMARY:
Purpose:

* evaluate the safety of Vorinostat.
* evaluate the effectiveness of Vorinostat in treating breast cancer
* evaluate how the study subject's body reacts to Vorinostat, how these reactions relate to the subject's genes, and whether protein changes in the subject blood may be used to predict how the subject's cancer will respond to Vorinostat

We hypothesize that Vorinostat, as a novel class of anti-cancer agents, may induce response in patients with recurrent or metastatic breast cancer who have been previously treated with anthracyclines and taxanes. In addition, we hypothesize that serum Vorinostat levels may correlate with clinical response and toxicities, and that Vorinostat may induce unique protein changes in the plasma in responding patients, and that these proteins may in turn be used as predictive biomarkers for treatment response.

DETAILED DESCRIPTION:
Breast cancer is sensitive to a range of chemotherapeutics agents, but despite initial sensitivity, resistance typically emerges, resulting in disease relapse or progression. Exploration of novel classes of agents in the treatment of breast cancer is therefore in urgent need. Vorinostat or SAHA, a potent inhibitor of histone deacetylase (HDAC) activity, represents a novel class of anti-cancer agents in early stages of development. Vorinostat is active in inducing differentiation, cell growth arrest, and/or apoptosis in a wide variety of transformed cells in culture, and has shown activity against breast cancer in cell lines and animal models. Exploratory pharmacokinetic analysis has demonstrated that oral Vorinostat has excellent bioavailability. Oral Vorinostat has been administered to more than 300 patients enrolled in completed or ongoing clinical studies. The maximum tolerated dose (MTD) is 400 mg q.d. or 200 mg b.i.d. continuously, or 300 mg b.i.d. x 3 consecutive days per week. Dose-limiting toxicities (DLT) are non-hematologic (anorexia, dehydration, diarrhea and fatigue), that resolve quickly once drug administration is interrupted. This study will evaluate the safety and efficacy of Vorinostat in breast cancer patients who have failed anthracyclines and taxanes, and if proven active, will add an important new class of agents to the treatment armamentarium of breast cancer. The study will be divided into 2 phases: phase I to determine the MTD in our population, starting with 400mg q.d. continuously, with progressive dose decrements in the event of DLT; and phase 2 to determine efficacy of Vorinostat at MTD in 12-37 evaluable patients. Correlative studies (pharmacokinetics, pharmacogenetics, plasma proteomics, tumor histone acetylation, genomics and proteomics) will be carried out to identify markers that will predict treatment response and/or toxicity to Vorinostat, to achieve the future goal of tailored therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Cytologically or histologically confirmed adenocarcinoma of the breast that is recurrent and/or metastatic
* Must have measurable disease as defined by RECIST criteria
* No more than 2 prior chemotherapy for recurrent and/or metastatic disease excluding neoadjuvant or adjuvant chemotherapy
* Previously received anthracycline- and taxane-containing chemotherapy for treatment of breast cancer in the neoadjuvant, adjuvant, or metastatic setting
* Must be able to swallow capsules
* Adequate bone marrow reserve and liver function
* Women in reproductive age group must agree to practice effective contraception during the entire study period unless documentation of infertility exists.

Key Exclusion Criteria:

* Prior treatment with any HDAC inhibitor. Patients who have received such agents for other indications, e.g. epilepsy, may enroll in the trial after a 30 day washout period.
* Known CNS involvement by tumor
* Concurrent use of oral retinoids or any vitamin A, other than a single multivitamin tablet daily
* Acute infection requiring intravenous antibiotics or antifungal agents,known HIV infection, active hepatitis B and/or hepatitis C infection
* Uncontrolled intercurrent illness
* Cancer other than breast cancer with the exception of basal cell carcinoma or disease that has been in remission for ≥5 years
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Clinical laboratory tests | Screening (Visit 1) and weekly during Cycle 1
  Laboratory tests will include the following: full blood count, albumin, alkaline phosphatase, total bilirubin, BUN, calcium, chloride, creatinine, glucose, LDH, potassium, total protein, AST, ALT, sodium and uric acid
Vital signs | Screening (Visit 1) and at subsequent visits
  Vital signs will include pulse, blood pressure, temperature, and respiration rate. Any treatment-emergent clinically significant vital sign abnormalities should be reported and followed as an adverse event.
Electrocardiograms | (Visit 1) and every 12 weekly while on treatment.
  ECG results will be reviewed by the investigator, and any treatment-emergent clinically significant ECG abnormality should be reported and followed as an adverse event.

SECONDARY OUTCOMES:
Vorinostat concentration in serum samples | Cycle 1 Day 1 (Week 1) and Cycle 1 Day 15 (Week 3)
  Vorinostat and its two metabolites SAHA-glucuronide and n-phenyl succinamic acid in human serum samples will be isolated by high throughput liquid chromatograph (HTLC) on-line extraction system.AUC, terminal elimination rate constant,total serum clearance (CL), volume of distribution (Vz) and bioavailability after oral administration will be calculated
Level of histone H3 acetylation | Baseline and 3 weeks after initiation of Vorinostat treatment
  10ml whole blood will be collected in heparinized tubes at baseline and 3 weeks after initiation of Vorinostat treatment, and centrifuged to obtain peripheral mononuclear cells. Histones will be isolated and acetylated histone H3 evaluated by Western blot analysis and enzyme linked immunosorbent assay (ELISA).
Known functional single nucleotide polymorphisms | prior to start of treatment
  Known functional single nucleotide polymorphisms (SNPs) of genes encoding for proteins that are relevant to the pharmacokinetic disposition and pharmacodynamics of Vorinostat will be characterized. More comprehensive genotyping using high-throughput sequencing techniques will be carried out in 'outliers' who have extreme pharmacokinetic parameters, or who experience exceptional toxicity or tumor response, to identify novel functional SNPs.
Baseline plasma protein profiles and changes in response to chemotherapy | baseline, on day 1 of each subsequent treatment cycle for the first 6 cycles, followed by 3 monthly until documented disease progression.
  Plasma proteomics studies using SELDI-MS with the Ciphergen technology will be collected serially to identify protein markers that are associated with Vorinostat response.
Tumor histone acetylation studies, genomics and proteomics studies (optional) | at baseline, and 3 weeks after initiation of Vorinostat treatment
  Tumor samples will be snap frozen in liquid nitrogen for subsequent RNA and protein extraction for tumor histone acetylation studies, gene expression studies and proteomic studies in an attempt to identify biomarkers that correlate with Vorinostat biological effects and clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin LEE, MBBS,MRCP, Study Chair — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore

REFERENCES:
- [Background] Munster PN, Troso-Sandoval T, Rosen N, Rifkind R, Marks PA, Richon VM. The histone deacetylase inhibitor suberoylanilide hydroxamic acid induces differentiation of human breast cancer cells. Cancer Res. 2001 Dec 1;61(23):8492-7. PMID 11731433
- [Background] Kelly WK, O'Connor OA, Krug LM, Chiao JH, Heaney M, Curley T, MacGregore-Cortelli B, Tong W, Secrist JP, Schwartz L, Richardson S, Chu E, Olgac S, Marks PA, Scher H, Richon VM. Phase I study of an oral histone deacetylase inhibitor, suberoylanilide hydroxamic acid, in patients with advanced cancer. J Clin Oncol. 2005 Jun 10;23(17):3923-31. doi: 10.1200/JCO.2005.14.167. Epub 2005 May 16. PMID 15897550